CLINICAL TRIAL: NCT00625963
Title: The Study of CT Scan and Echocardiogram Parameters in Patients With Pulmonary Hypertension With Regards to Hemodynamics, Sleep Studies, and Various Laboratory Markers.
Brief Title: The Study Of CT Scans and Echo Parameters in Patients With PAH
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 07.060
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension;; ILD;; CT Imaging;; Echocardiogram;; Hemodynamic measurements of RHC.; Pulmonary Function Tests
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I,A: I=Pulmonary Hypertension Patients A=ILD patients with Pulmonary Hypertension Patients

SUMMARY:
Current standard of the diagnosis and monitoring of PHNT requiring combination of invasive and non-invasive tests. The goal of the study is to correlate data from CT scans, echocardiograms, right heart catheterization, PFTs, sleep studies, and perfusion scans. The ultimate goal is to determine patterns of the PAH disease processes.

DETAILED DESCRIPTION:
The goal of our study is to correlate data from various non-invasive tests such as commuted tomography (CT) imaging, echocardiogram, Pulmonary Function Tests, and other laboratory tests along with hemodynamic measurements from Right Heart Catheterizations in these ILD patients with Pulmonary Hypertension, as well as all other pulmonary hypertension. The ultimate goal is to determine patterns of the PAH disease processes, as well as define optimal diagnostic modalities including in-hospital verses outpatient studies.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Hypertension;
* ILD with Pulmonary Hypertension

Exclusion Criteria:

* NON-PH

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary Arterial Hypertension; Idiopathic Lung Disease
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The Study Of CT Scans and Echo Parameters in Patients With PAH | All data has been previously collected.
  Correlation of Pulmonary artery diameter as measured by CT scan and Pulmonary artery systolic pressure as measured by Echocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Arunabh Talwar, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore-Long Island Jewish Health System, New Hyde Park, New York, United States